CLINICAL TRIAL: NCT06920394
Title: Functionality of Lower Limbs in Patients Who Have Undergone Knee Meniscectomy. A Multicenter Ambispective Cohort Study
Brief Title: Functionality of Lower Limbs in Patients Who Have Undergone Knee Meniscectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: FunctMenisc
Record Dates: First submitted 2025-04-01; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Meniscectomy Sequelae
Keywords: Knee meniscectomy; Functionality; Range of movement; Pain intensity; Kinesiophobia
MeSH Terms: conditions — Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients will be recruited from the Fisiomaturana and Fisialty centers. The primary variable of the study will be functionality, with the prescription of a post-surgical physiotherapy treatment being the dependent variable. The secondary variables, estimated as modifying or confounding, will be range of motion, pain intensity and kinesiophobia.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — In the present study, no intervention will be carried out, and only the patients recruited will complete the questionnaires set out below.

SUMMARY:
Introduction. Meniscal lesions are common and are associated with the development of osteoarthritis of the knee. Work activities that cause mechanical stress can lead to acute or chronic injuries. The surgical treatment for this injury is meniscectomy. Physiotherapy is a widely accepted first-line treatment for patients with meniscus tears.

Objective. To assess the clinical and functional status of patients who have undergone meniscus surgery with and without post-surgical physiotherapy.

Material and method. Multicenter ambispective cohort study. 89 patients who have undergone meniscectomy will be recruited. The primary variable of the study will be functionality (Time Up & Go), with the prescription of a post-surgical physiotherapy treatment being the dependent variable. The secondary variables, estimated as modifying or confounding, will be range of motion (goniometry), pain intensity (visual analog scale) and kinesiophobia (Tampa scale).

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 20 to 65
* Of both sexes
* With previous meniscectomy surgery in one of the two knees in the last 5 years
* Who sign the informed consent document.

Exclusion Criteria:

* Patients who require technical aids for walking
* Dependent patients for carrying out activities of daily living
* Patients over 65 years of age
* Patients with cognitive impairments that prevent understanding of tests and evaluations

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with previous meniscectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of knee functionality | Screening visit
  To assess knee functionality we will use the Time Up & Go instrument. This test consists of getting up from a chair, walking three meters around an obstacle and returning to the starting position. This tool is closely related to the risk of falls. The unit of measurement is time, where the lower the mark, the better the functionality.

SECONDARY OUTCOMES:
Assessment of range of knee motion | Screening visit
  The range of knee motion will be assessed using a goniometer. The fixed arm will be placed between the center of the greater trochanter and the lateral epicondyle of the femur, while the movable arm will be placed on the axis of the tibia between the lateral femoral epicondyle and the center of the lateral malleolus. During the evaluation, each patient will be asked to perform maximum active knee flexion and extension. The unit of measurement is the maximum range of motion measured in degrees, where the higher the graduation, the greater the range of motion.
Assessment of pain perception | Screening visit
  Pain perception will be measured using a visual analog scale. This measuring instrument quantifies pain according to the patient's subjective perception on a scale of 0 to 10, where 0 indicates the absence of pain and 10 the maximum pain perceived by the patient.
Assessment of Kinesiophobia | Screening visit
  Kinesiophobia (fear of movement) will be measured using the Tampa Scale (TSK-11). This scale consists of 11 questions scored from 1 "strongly disagree" to 4 "strongly agree". The range of scores is from 11 to 44 points, where a higher score indicates greater fear of movement on the part of the respondent.

OTHER OUTCOMES:
Assessment of the time elapsed since the surgical intervention | Screening visit
  The main clinical variables will be measured: date of the surgical procedure and date of evaluation (in DD/MM/YYYY format; to calculate the elapsed time, in days)
Assessment of the patient's weight at the time of the study | Screening visit
  The anthropometric variables of weight (measured in kg)
Measurement of the patient's age at the time of the study | Screening visit
  The sociodemographic variables age (in whole months) will be measured
Assessment of the patient's height at the time of the study | Screening visit
  The anthropometric variable height (measured in cm)
Assessment of the patient's gender at the time of the study | Screening visit
  The sociodemographic variable gender (male/female) will be measured
Assessment of the patient's type of work at the time of the study | Screening visit
  The sociodemographic variable type of work (sedentary/active) will be measured. This evaluation will be based on whether the work is office work or at least 4 hours/day sitting.
Measurement of the patient's level of physical activity before and after surgery | Screening visit
  The variable physical exercise before and after meniscectomy will be measured (dichotomous answers: yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided